CLINICAL TRIAL: NCT02018185
Title: The Efficacy of Deep Repetitive Transcranial Magnetic Stimulation in Treatment of Obsessive Compulsive Disorder, a Double Blind Randomized Clinical Trial
Brief Title: Study of Magnetic Brain Stimulation in Treatment of Obsessive Compulsive Disorder
Acronym: rTMS
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment has been suspended in order to perform interim data analysis.
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Medical Service Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B2013:144
Record Dates: First submitted 2013-12-10; First posted 2013-12-23 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial Magnetic Stimulation (Active Comparator): Transcranial Magnetic Stimulation
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham Transcranial Magnetic Stimulation
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — A non-invasive method for brain stimulation
  Arms: Transcranial Magnetic Stimulation
Device: Sham Transcranial Magnetic Stimulation — Sham stimulation of the brain.
  Arms: Sham rTMS

SUMMARY:
In a preliminary pilot study, the investigators tested the efficacy of rTMS over the medial prefrontal cortex in symptom profiles of obsessive compulsive disorder (OCD) patients. This study revealed considerable benefit in using rTMS for the treatment of OCD.

In the current proposal, in a randomized clinical trial, the investigators aim to further evaluate the efficacy of rTMS in OCD in a larger sample size and for a longer period. Studies into the efficacy of rTMS in other psychiatric disorders such as depression have consistently shown that extension of the treatment to four weeks significantly increased the effect size. In the pilot study, the investigators applied rTMS for only two weeks. Although all patients consistently showed improvement in their symptoms, none of them showed complete remission of their OCD. Here, the investigators hypothesize that longer duration of rTMS treatment will have greater benefit in OCD symptom reduction.

DETAILED DESCRIPTION:
The purpose of study is to examine the efficacy of rTMS over the medial prefrontal cortex in the treatment of OCD.

rTMS will be provided to OCD patients in a randomized double blind controlled setting, and the investigators hypothesize that in this setting the treatment group would still show significant improvement in OCD symptoms as compared to the sham group.

rTMS will be applied for four weeks on OCD patients and the investigators will assess improvement after four weeks of rTMS. The investigators hypothesize that patients will show significantly greater improvement after four weeks of rTMS vs. two weeks of rTMS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed obsessive compulsive disorder
* Not currently receiving cognitive behavioural therapy
* Not currently on any medication or only taking one selective serotonin reuptake inhibitor (SSRI)

Exclusion Criteria:

* History of psychotic episodes
* History of neurological illness
* Previous head injury
* Active alcohol or substance abuse
* History of seizure disorders
* Currently pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in obsessive and compulsive symptom severity (Yale-Brown Obsessive Compulsive Scale) | Recordings: baseline; after two weeks of rTMS; after four weeks of rTMS; monthly for three months following the last session of rTMS

CONTACTS AND LOCATIONS:
Locations (1):
- St. Boniface Hospital, Winnipeg, Manitoba, Canada